CLINICAL TRIAL: NCT01213004
Title: Evaluation of Respiratory Motion-Corrected Cone-Beam CT in Radiation Treatment of Thoracic and Abdominal Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-146
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Gastric Cancer; Lung Cancer
Keywords: gastro-esophageal junction; lung; abdominal; cone-beam CT (CBCT); 10-146
MeSH Terms: conditions — Stomach Neoplasms; Lung Neoplasms

ARMS (2):
- thoracic (study group 1) malignancies (Experimental): On the same day as the CBCT scans and treatment session, patients will receive a research-only respiration correlated CT (RCCT scan), for calculating motion-corrected CBCT. The localization accuracy of motion-corrected CBCT using same-day RCCT will be compared to that using the standard RCCT from simulation.
  Interventions: Procedure: respiration correlated CT scan
- abdominal (study group 2) malignancies (Experimental): On the same day as the CBCT scans and treatment session, patients will receive a research-only respiration correlated CT (RCCT scan), for calculating motion-corrected CBCT. The localization accuracy of motion-corrected CBCT using same-day RCCT will be compared to that using the standard RCCT from simulation.
  Interventions: Procedure: respiration correlated CT scan

INTERVENTIONS:
Procedure: respiration correlated CT scan — Thoracic malignancies (study group 1): Patients to be treated for gastro-esophageal junction (GEJ) malignancy undergo an implantation procedure of two or three radiopaque markers several days prior to treatment simulation, which are used to correct patient position at treatment. At treatment simulation, patients receive a standard CT scan followed by an RCCT scan. In cases of GEJ malignancy, oral contrast is administered prior to the standard CT scan; this is done at the treating physician's discretion. The standard CT is used to design the radiation treatment plan, where as the RCCT is used to define a volume that encompasses the motion extent of the tumor with breathing and is transferred to the standard CT.
  Arms: thoracic (study group 1) malignancies
Procedure: respiration correlated CT scan — Abdominal malignancies (study group 2): Patients undergo an implantation procedure of two or three radiopaque markers several days prior to treatment simulation. At treatment simulation, patients receive a standard CT scan followed by an RCCT scan. Intravenous contrast is administered prior to the standard CT; this is done at the treating physician's discretion.
  Arms: abdominal (study group 2) malignancies

SUMMARY:
Tumors must be seen clearly on CT scan to be radiated completely and safely. Breathing causes tumors to move. If the tumor moves during breathing, it can look blurred on the CT scan. This makes it difficult to see on CT scan. The investigators wish to investigate whether a new computer method makes tumors less blurry and easier to see on CT scan. Cone-beam CT is a type of CT scanner attached to the radiation treatment machine that produces 3D images of the patient. Since your tumor can move because of your normal breathing, it is often blurry and difficult to see accurately in a standard cone-beam CT scan. The investigators intend to use a computer method which processes the cone-beam CT data in a way that reduces the blurring and makes the tumor easier to see.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic proof of a thoracic or abdominal malignancy, confirmed at MSKCC and suitable for radiation therapy, in order to be eligible for this study. Thoracic malignancies (study group 1) include those in lung and gastro-esophageal junction. Abdominal malignancies (study group 2) include those in liver and pancreas. Patients having both thoracic and abdominal malignancies will be placed in only one of the study groups, because the limited field-of-view of the CBCT precludes imaging of both malignancies in the same scan. Patients must be older than 18 years of age
* At least part of the tumor must be visible as observed in a diagnostic or planning CT. The tumor must exhibit at least 5 mm motion from respiration as observed in the respiration-correlated CT (RCCT) at simulation. The RCCT scan must be interpretable and not exhibit excessive motion artifacts caused by irregular patient breathing.
* Patients must have Karnofsky Performance Status ≥ 70%

Exclusion Criteria:

* Mesothelioma and other tumors of the pleura
* Pregnant Women
* Allergic to iodine or intravenous contrast agent (applies only to patients with a pancreas or liver malignancy)
* Renal impairment due to the use of a contrast agent
* Patients with pacemakers and defibrillators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
To determine whether motion-corrected cone-beam CT (CBCT) improves the localization accuracy | 2 years
  of thoracic tumors (evaluated using study group 1) and organs-at-risk (evaluated using study group 2) relative to the standard cone-beam CT procedure.
To determine whether motion-corrected cone-beam CT (CBCT) can visualize and localize abdominal tumors using intravenous contrast enhancement. | 2 years
  (evaluated using study group 2).

SECONDARY OUTCOMES:
To determine whether motion-corrected cone-beam CT (CBCT) derived from a respiration correlated CT (RCCT) scan on the same day improves localization accuracy | 2 years
  for thoracic tumors (evaluated using study group 1) and organs-at-risk (evaluated using study group 2), relative to motion-corrected CBCT derived from a prior RCCT scan at patient's simulation.
To determine whether tumor and organ-at-risk positions localized in cone-beam CT (CBCT) | 2 years
  prior to treatment remain constant throughout the treatment fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Gikas Mageras, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm